CLINICAL TRIAL: NCT06103825
Title: A Double-blind, Placebo-controlled, Randomized, Parallel-group, Multicenter Study to Evaluate the Efficacy and Safety of the Treatment with Solriamfetol in Excessive Daytime Sleepiness (EDS) in Patients with Obstructive Sleep Apnea Syndrome (OSA) with a 12-week Treatment Period
Brief Title: A Twelve-week, Double-blind, Placebo-controlled, Randomized, Parallel-group, Multicenter Study to Evaluate the Efficacy and Safety of Solriamfetol in the Treatment of Excessive Daytime Sleepiness (EDS) in Patients with Obstructive Sleep Apnea (OSA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ignis Therapeutics (Suzhou) Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IGN-B0301-03
Record Dates: First submitted 2023-09-27; First posted 2023-10-27 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2024-10

CONDITIONS: Sleep Apnea, Obstructive; Excessive Daytime Sleepiness
MeSH Terms: conditions — Sleep Apnea, Obstructive; Disorders of Excessive Somnolence | interventions — solriamfetol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Strengths of solriamfetol (JZP-110) strengths: 37.5 mg，75 mg, 150 mg (Experimental): subject will first enter a 2-week Titration Phase, during which the initial dose will be 37.5mg. The dose will be increased from 37.5mg QD to 75mg QD after 3 days, and then to 150mg QD at the first day of the second week if well-tolerated. subjects will then enter the 10-week Maintenance Phase on 150mg QD if well-tolerated.
  If a subject tolerability issues after titration up to 150mg at the second week, the dose can be reduced to 75mg QD following instructions of the investigators. This subject will then enter the 10-week Maintenance Phase on 75mg QD.
  If a subject experiences tolerability issues after titration up to 75mg at the first week, the dose can be reduced to 37.5mg QD following instructions of the investigators. The dose will be increased to 75mg QD again at the first day of the second week. Subject will then enter the 10-week Maintenance Phase on 75mg QD if well-tolerated.
  All subjects should be maintained on either 75mg QD or 150mg QD during the Maintenance Phase.
  Interventions: Drug: Solriamfetol
- matching Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Solriamfetol — solriamfetol : QD，PO，Day 1-Day 84；
  Arms: Strengths of solriamfetol (JZP-110) strengths: 37.5 mg，75 mg, 150 mg
Drug: Placebo — Placebo :QD，PO，Day 1-Day 84
  Arms: matching Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of 12-week solriamfetol administration in the treatment of EDS in patients with OSA from China, using a randomized, double-blind, placebo-controlled, multi-center, parallel-design.

ELIGIBILITY:
Inclusion criteria:

1. Male or female between 18 to 75 years of age, inclusive.
2. Diagnosis of OSA according to the International Classification of Sleep Disorders, 3rd edition (ICSD-3) criteria.
3. Patients with OSA may be considered for enrollment if they meet one of the following criteria:

   1. Use of a primary therapy for OSA (i.e., positive airway pressure (PAP), oral pressure therapy, oral appliance, or upper airway stimulator) on at least 1 night per week, or
   2. History of at least 1 month of an attempt to use one or more primary OSA therapies with at least one documented adjustment that was made in an attempt to optimize the primary OSA therapy, or participants who have never used and refuse to use a primary OSA therapy, or
   3. History of a surgical intervention intended to treat OSA symptoms.
4. A stable level of compliance with a primary OSA therapy for at least 1 month prior to the baseline visit as follows:

   1. A stable level of use of a primary OSA therapy, or
   2. A lack of use of a primary OSA therapy either following a history of attempted use, or have never used before, or
   3. A history of a surgical intervention intended to treat OSA symptoms.
5. Baseline ESS score no less than 10 points (≥ 10 points).
6. Baseline MWT mean sleep latency < 30 minutes (documented by the mean of the first four 40-minute trials of the MWTs).
7. Usual nightly total sleep time of at least 6 hours (≥ 6 hours).
8. Body mass index (BMI) from18 kg/m2 to < 45 kg/m2.
9. Female participants must have negative pregnancy test results at the screening and baseline visits; all participants must consent to use a medically acceptable method of contraception throughout the entire study period and for 30 days after the study is completed.
10. Willing and able to provide written informed consent, willing and able to comply with the study protocol (i.e., must be able to understand and complete the study questionnaires and scales, comply with the visit schedule and prescribed dosage regimens).
11. Determined by the investigator to be medically stable as assessed by medical history, physical examination, laboratory and electrocardiogram test results and review of concomitant medications.

Exclusion criteria：

1. Female participants who are pregnant or lactating.
2. Usual bedtime later than 1 a.m. (01:00).
3. Occupation requiring nighttime shift work or variable shift work.
4. Any other clinically relevant medical, behavioral, or psychiatric disorders other than OSA that is associated with excessive sleepiness.
5. History or presence of bipolar disorder, bipolar related disorders, schizophrenia, schizophrenia spectrum disorder, or other psychotic disorders according to DSM-5 criteria, or presence of significant suicidality.
6. History or presence of any acutely unstable medical condition, behavioral or cognitive impairment, or any medical condition or surgical history that could affect the safety of the participant or interfere with study efficacy, safety and PK assessments, or the ability of the participant to complete the study per the judgment of the investigator.
7. History of the bariatric surgery within the past year or a history of any gastric bypass procedure.
8. Presence of renal impairment or calculated creatinine clearance less than 60 mL/min at screening, which is calculated using the following formula: CLcr (mL/min) = (140 - age [years]) x body weight (kg) x (0.85, if female))/(72 x serum creatinine value [mg/dL]), if serum creatinine is expressed in µmol/L, the value should be divided by 88.4 to convert µmol/L to mg/dL.
9. Clinically significant ECG abnormality in the opinion of the investigator would preclude participation in the study.
10. Presence of significant cardiovascular disease at screening, including but not limited to: myocardial infarction within the past year, unstable angina pectoris, symptomatic congestive heart failure [(American College of Cardiology/American Heart Association (ACC/AHA) Stage C or D)], revascularization procedures within the past year, ventricular cardiac arrhythmia requiring an automatic implantable cardioverter defibrillator (AICD) or medication therapy, uncontrolled hypertension, systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 95 mmHg (at Screening, or across Baseline measures according to protocol specifications), or any significant cardiovascular condition that in the investigator's opinion may jeopardize participant's safety in the study.
11. Laboratory value(s) outside the laboratory reference range that are considered to be clinically significant and may affect the safety of the participant per the judgment of the investigator (including clinical chemistry, hematology, and urinalysis) (Note: Screening labs may be repeated once).
12. Excessive caffeine use one week prior to the baseline assessments, or anticipated excess caffeine use during the study, defined as greater than 600 mg caffeine per day (>600 mg/day).
13. Use of any over-the-counter (OTC) or prescription medications that could affect the evaluation of excessive sleepiness within a time period prior to the baseline visit corresponding to at least five half-lives of the drug(s) or planned use of such drug(s) at some point throughout the duration of the study. Examples of excluded medications include OTC sleep aids or stimulants (e.g., pseudoephedrine), methylphenidate, amphetamines, modafinil, 2-acetamide, sodium oxybate, pemoline, trazodone, hypnotics, benzodiazepines, barbiturates, and opioids, and any traditional Chinese medicine that may affect sleep. Medications should be discontinued such that the participant has returned to his/her baseline level of daytime sleepiness at least 7 days prior to the baseline visit, in the opinion of the investigator.
14. Use of a monoamine oxidase inhibitor (MAOI) in the past 14 days or five half-lives (whichever is longer) prior to the baseline visit or plans to use an MAOI during the study.
15. Received an investigational drug or device in the past 30 days or five half-lives (whichever is longer) prior to the baseline visit, or plans to use an investigational drug (other than the investigational drug) or investigational medical devices during the study
16. Previous exposure to or participation in a clinical trial of solriamfetol.
17. Current or past (within the past 2 years prior to screening) diagnosis of a moderate or severe substance use disorders according to DSM-5 criteria or seeking treatment for a substance related disorder.
18. Nicotine dependence that has an effect on sleep (e.g., a participant who routinely awakened at night to smoke).
19. Urine drug screen positive for an illicit drug of abuse (including cannabinoids) at screening or at any point throughout the duration of the study, except for a prescriped drug (e.g., amphetamines) at screening.
20. History of phenylketonuria (PKU) or history of hypersensitivity to phenylalanine-derived products.
21. Vaccination within 31 days prior to the baseline visit or a plan for vaccination during the study.
22. Any other conditions that are not in line with the rights and interests of the participants or would preclude participation in the study as judged by the investigator.
23. Human Immunodeficiency Virus (HIV) or syphilis positive at screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-08-19 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of solriamfetol compared to placebo among patients with OSA in change from baseline to Week 12 in the mean MWT sleep latency (minutes, (determined from the first four 40-minute trials of the MWT) | From enrollment to the end of treatment at 12 weeks
  Change from baseline in mean MWT sleep latency (minutes, determined from the first four 40-minute trials of the MWT) to Week 12
To evaluate the effect of solriamfetol compared to placebo among patients with OSA in change from baseline to Week 12 in ESS scores | From enrollment to the end of treatment at 12 weeks
  Change from baseline in ESS total score to Week 12 Epworth Sleepiness Scale (ESS): ESS score ranges from 0 to 24 (inclusive), with higher score denoting greater degrees of sleepiness

SECONDARY OUTCOMES:
Key Secondary Study Objective: To compare treatment with solriamfetol versus placebo on the percentage of participants reported as improved (minimally, much, very much) in PGIc at Week 12 among patients with OSA | From enrollment to the end of treatment at 12 weeks
  Percentage of participants with improved PGIc at Week 12
Other Secondary Study Objective 1:To evaluate the effect of solriamfetol compared to placebo among patients with OSA in change from baseline to Week 2 and Week 5 in the mean MWT sleep latency | From enrollment to the end of treatment at the 2- and 5-week
  Changes from baseline in MWT at the end of the Week 2 and Week 5 are defined as: mean sleep latency at the end of the Week 2 and Week 5 (determined from the first four 40-minute trials of the MWTs) minus the baseline measurement (minutes)
Other Secondary Study Objective 2: To evaluate the effect of solriamfetol compared to placebo among patients with OSA in change from baseline to Week 2, 5 and 8 in ESS score | From enrollment to the end of treatment at the 2- ,5- and 8-week
  Changes from baseline in ESS scores at the end of Week 2, 5 and 8 are defined as: ESS total scores at the end of Week 2, 5 and 8 minus baseline values Epworth Sleepiness Scale (ESS): ESS score ranges from 0 to 24 (inclusive), with higher score denoting greater degrees of sleepiness
Other Secondary Study Objective 3: To compare treatment with solriamfetol versus placebo on the percentage of participants reported as improved (minimally, much, very much) in PGIc at Week 2, 5 and 8 among patients with OSA | From enrollment to the end of treatment at the 2- ,5- and 8-week
  The percentages of participants reported as improved (minimally, much, very much) in PGIc at Week 2, 5 and 8 are defined as the percentages calculated by dividing the number of participants reported as improved in PGIc by the total number of participants in the each treatment group at Week 2, 5 and 8
Other Secondary Study Objective 4: To compare treatment with solriamfetol versus placebo on the percentage of participants rated as improved (minimally, much, very much) in CGIc at Week 12 among patients with OSA | From enrollment to the end of treatment at 12 weeks
  The percentage of participants rated as improved (minimally, much, very much) in CGIc at the end of Week 12 is defined as the percentage calculated by dividing the number of participants who have achieve improvement (minimally, much, very much) in CGIc by the total number of participants in each treatment group at Week 12
Other Secondary Study Objective 5: To compare treatment with solriamfetol versus placebo on the percentage of participants rated as improved (minimally, much, very much) in CGIc at Week 2, 5 and 8 among patients with OSA | From enrollment to the end of treatment at the 2- ,5- and 8-week
  The percentage of participants rated as improved (minimally, much, very much) in CGIc at the end of Week 12 is defined as the percentage calculated by dividing the number of participants who have achieve improvement (minimally, much, very much) in CGIc by the total number of participants in each treatment group at Week 2, 5 and 8
Other Secondary Study Objective 6: To compare the efficacy of solriamfetol versus placebo throughout the day in sleep latency for each of the 5 MWT trials | From enrollment to the end of treatment at 12 weeks
  Changes of the efficacy throughout the day in MWT: changes in sleep latency for each of the 5 MWTs (minutes)

CONTACTS AND LOCATIONS:
Locations (26):
- China (26):
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - Beijing TianTan Hospital Capital Medical University, Beijing
  - China-Japan friendship Hospital, Beijing
  - Peking University Sixth Hospital, Beijing
  - XuanWu Hospital Capital Medical University, Beijing
  - The first hospital of Jilin University, Changchun
  - Xiangya Hospital Central South University, Changsha
  - ChongQing University three gorges Hospital, Chongqing
  - The Hospital Group of the First Affiliated Hospital of CQMU, Chongqing
  - GanSU Provincial Hospital, Gansu
  - The first affiliated hospital of Guangzhou Medical University, Guangzhou
  - The first affiliated hospital of JiNan University, Guangzhou
  - Hangzhou seventh People's Hospital, Hangzhou
  - The first hospital of Hebei Medical University, Hebei
  - Huai'an First People's Hospital, Huai'an
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - The Fitst Affiliated Hospital of NingBo University, Ningbo
  - ShanDong Provincial QianFoShan Hospital, Shandong
  - HuaShan Hospital FuDan University, Shanghai
  - First hospital of ShanXi Medical University, Shanxi
  - Second hospital of Shanxi Medical University, Shanxi
  - ShenZhen People's Hospital, Shenzhen
  - West China fourth Hospital Sichuan University, Sichuan
  - The Second Affiliated Hospital of Suzhou University, Suzhou
  - Yan'an University Xianyang Hospital, Xianyang
  - The First People's Hospital of YunNan Province, Yunnan

REFERENCES:
- [Derived] Cheng H, Deng L, Meng Z, Zhang W, Chen T, Chen R, Tang S, Lv Y, Su X, Liu Z, Zhang X, Wang X, Mao H, Zhang N, Yu H, Pan J, Xie Y, Tang J, Yin S, Wang Z, Tong M, Zhan S, Wang C, Wang B, Zhang W, Mi W, Lu L. Efficacy and Safety of Solriamfetol on Excessive Daytime Sleepiness Associated with Obstructive Sleep Apnea in China: A Phase 3, Multicenter, Double-Blind, Placebo-Controlled Randomized Clinical Trial. CNS Drugs. 2026 Jan;40(1):83-98. doi: 10.1007/s40263-025-01232-1. Epub 2025 Oct 23. PMID 41128833